CLINICAL TRIAL: NCT01538576
Title: Special Survey for Paediatric Subjects
Brief Title: Paediatric Subjects - Special Survey
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1942
Record Dates: First submitted 2012-02-15; First posted 2012-02-24 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin aspart users
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Prescribed by the physicians as a result of normal clinical practice

SUMMARY:
This study is conducted in Japan. The aim of this study is to collect safety and efficacy data when using insulin aspart in children with diabetes under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diabetes requiring insulin therapy

Exclusion Criteria:

* Subjects who had treatment history of insulin aspart

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients under 15 years of age with diabetes requiring insulin therapy with no treatment history of insulin aspart (NovoRapid®)
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2003-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Response rate assessed by the investigator: Ability or failure to achieve expected glycaemic control | Year 1
HbA1c (glycosylated haemoglobin) | Year 1

SECONDARY OUTCOMES:
Hypoglycaemic events | Year 1
Adverse Events | Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com